CLINICAL TRIAL: NCT06704646
Title: Predictors of One-Year Mortality After Curative Surgery in Patients Aged 80 Years or Older With Non-Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202003045RINB
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Geriatrics
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients passed away within one year: Records their age, gender, preoperative comorbidities, and calculated their Charlson comorbidity index. We also collected information on tumor location, serum levels of carcinoembryonic antigen (CEA), preoperative clinical TNM staging, and postoperative pathological TNM staging
  Interventions: Procedure: Curative intent surgery
- Patient survived the first post-operative year: Records their age, gender, preoperative comorbidities, and calculated their Charlson comorbidity index. We also collected information on tumor location, serum levels of carcinoembryonic antigen (CEA), preoperative clinical TNM staging, and postoperative pathological TNM staging
  Interventions: Procedure: Curative intent surgery

INTERVENTIONS:
Procedure: Curative intent surgery — Curative intent surgery means that surgeons intend to perform R0 resection.

SUMMARY:
The aim of this study is to determine which preoperative factors are associated with one-year postoperative mortality in patients aged ≥80 years undergoing curative surgery and compare outcomes between patients with or without risk factors.

DETAILED DESCRIPTION:
Colorectal cancer is common among older adults, and with the aging global population, the number of elderly individuals diagnosed with this condition continues to rise. Current treatment guidelines identify surgery as the primary approach for managing non-metastatic colorectal cancer. Previous studies have shown that factors like advanced age, frailty, comorbidities, and nutritional status can predict surgical outcomes. However, in patients over 80 years old with non-metastatic colorectal cancer, questions remain regarding the definition of advanced age and frailty, the applicability of existing assessment tools to this specific group, and the determination of optimal cut-off values, all of which require further validation. Furthermore, there is a shortage of effective outpatient screening tools to identify vulnerable patients and provide reliable guidance for predicting postoperative survival. Therefore, the aim of this study is to determine which preoperative factors are associated with one-year postoperative mortality in patients aged ≥80 years undergoing curative surgery and compare outcomes between patients with or without risk factors.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥80 years with stages I-III colorectal cancer who underwent tumor resection from January 2014 to January 2019

Exclusion Criteria:

Patients undergoing procedure without colectomy, or tumor excised by transanal method were excluded from this study

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This retrospective study was performed at National Taiwan University hospital. Patients aged ≥80 years with stages I-III colorectal cancer who underwent tumor resection from January 2014 to January 2019, and they were followed up until December 31, 2020. Patients undergoing procedure without colectomy, or tumor excised by transanal method were excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Preoperative factors associated with one-year postoperative mortality | From operation to one year after the surgery
  Univariate and multivariable logistic regression analysis were performed to identify preoperative factors associated with one-year postoperative mortality.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keum N, Giovannucci E. Global burden of colorectal cancer: emerging trends, risk factors and prevention strategies. Nat Rev Gastroenterol Hepatol. 2019 Dec;16(12):713-732. doi: 10.1038/s41575-019-0189-8. Epub 2019 Aug 27. PMID 31455888
- [Background] Chen B, Yu W, Ma Y, Xu P, Yao Q, Sun Q, Ren J, Wang D. Evaluation of the safety and efficacy of perform enterectomy in colorectal cancer patients aged 80 or older. A meta-analysis and a systematic review. Int J Colorectal Dis. 2023 Jul 3;38(1):185. doi: 10.1007/s00384-023-04461-2. PMID 37395836
- [Background] Dekker JW, van den Broek CB, Bastiaannet E, van de Geest LG, Tollenaar RA, Liefers GJ. Importance of the first postoperative year in the prognosis of elderly colorectal cancer patients. Ann Surg Oncol. 2011 Jun;18(6):1533-9. doi: 10.1245/s10434-011-1671-x. Epub 2011 Mar 29. PMID 21445672